CLINICAL TRIAL: NCT06305117
Title: VRtuose (Virtual RealiTy and mUsic in the Oncology SEtting) : A Single-centre Feasibility Study Evaluating a Strategy Combining Virtual Reality and Music to Improve Quality of Life in Breast Cancer Patients Undergoing Chemotherapy
Brief Title: Virtual RealiTy and mUsic in the Oncology SEtting - Phase 1
Acronym: VRtuose1
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: International Agency for Research on Cancer (Other)
Collaborators: Centre Leon Berard (Other)
Responsible Party: Principal Investigator, Pauline Boucheron, Postdoctoral scientist, International Agency for Research on Cancer
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: PP202304-37-1; 101227 (Other Grant/Funding Number: Association Ruban Rose)
Record Dates: First submitted 2024-02-22; First posted 2024-03-12 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2025-02

CONDITIONS: Breast Cancer
Keywords: quality of life; virtual reality; music; feasibility study
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Participants (Experimental): As this is a feasibility study, all patients included in this study will be offered the intervention.
  Interventions: Other: Distraction strategy

INTERVENTIONS:
Other: Distraction strategy — Distraction strategy combining the use of virtual reality and music

SUMMARY:
The VRtuose (Virtual RealiTy and mUsic in the Oncology Setting) project aims to evaluate the feasibility of implementing in day patient chemotherapy units a distraction strategy combining virtual reality (VR) and music which fits the needs of both breast cancer patients and healthcare providers (i.e., strategy administrators), and to evaluate its impact on patients' (i) perceived anxiety and pain during chemotherapy sessions, (ii) nausea/vomiting and mood disturbances in between chemotherapy sessions, and (iii) quality of life.

The present project is a non-randomized non-controlled prospective monocentric feasibility study which will focus on evaluating the feasibility of implementing the strategy in the target population and setting.

In the case that implementation of a distraction strategy combining virtual reality and music to improve quality of life of breast cancer patients during chemotherapy is deemed feasible, the efficacy of using this strategy to improve patients' experience of chemotherapy and long-term quality of life will be evaluated in a future randomized controlled trial informed and optimized by the results of the present work.

DETAILED DESCRIPTION:
VRtuose (phase 1) is a non-randomized, single-centre, prospective, feasibility study conducted in the day patient chemotherapy unit of the Centre Léon Bérard in Lyon. This study will include women diagnosed with breast cancer who are receiving or are planned to receive any chemotherapy regimen. As this is a feasibility study, there will be no control group and all participants will be offered the intervention.

The intervention will be implemented from the first chemotherapy session onwards until it has been offered at four distinct chemotherapy sessions or until the end of patients' chemotherapy course if it is ended earlier. The intervention will be offered in addition to the standard of care at the study hospital.

All women with breast cancer who are about to start or who have started chemotherapy will be considered for inclusion in the study. All participants will be offered the distraction strategy for four consecutive chemotherapy sessions spanning over their chemotherapy course (i.e., from the first session onwards) whenever the strategy is available for use.

The intervention will be characterised by a strategy combining immersive virtual reality and music delivered during chemotherapy sessions to breast cancer patients by trained oncology nurses. Different immersive environments and of music will be available to the choice of the patient. From the first chemotherapy session onwards, patients will be offered by oncology nurses to use the distraction strategy during their chemotherapy session. Patients who are willing to use the strategy will have the possibility to choose the content of the strategy and to use it for the duration of their choice. Patients will be followed up from recruitment until they have been offered four times to use the strategy (or until the end of their chemotherapy course if it ends earlier).

This study will assess the feasibility to implement such a strategy into a day-hospital chemotherapy unit at a major oncology centre, and will therefore collect information on feasibility, acceptability and tolerability outcomes of using the strategy in this context. The efficacy of the strategy to improve patients' quality of life will not be evaluated in this study.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis of breast cancer;
* Any disease stage;
* Patient must be receiving (i.e., with at least 4 remaining cures) or about to start palliative or curative neoadjuvant or adjuvant chemotherapy for their breast cancer at Centre Léon Bérard;
* Willingness and ability to comply with the study requirements;
* Patient must be covered by a medical insurance;
* Patient must understand, speak, read and write French.

Exclusion Criteria:

* History of condition contraindicating the use of virtual reality (e.g., epilepsy, severe motion sickness);
* Brain metastases;
* Any medical or psychosocial condition that would compromise the patient's compliance to the study procedures or would likely interfere with the completion of Patient-Reported Outcomes;
* Patients under tutorship or curatorship;
* Patients already included in another clinical trial ongoing at Centre Léon Bérard.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-11-20 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Patients' acceptance rate regarding the use of the distraction strategy. | Through study completion, an average of 8 months.
  Average of the number of times the strategy is used by each patient out of the number of chemotherapy cures it is offered to each patient.

SECONDARY OUTCOMES:
Accessibility of the strategy | Through study completion, an average of 8 months.
  Percentage of chemotherapy sessions when strategy administrators offer patients to use the strategy.
Duration of use of the strategy by patients | Through study completion, an average of 8 months.
  Time elapsed in between start of the first video and end of the last video watched by the participant.
Type of video content chosen by participants | Through study completion, an average of 8 months.
  Measured using a questionnaire
Type of music content chosen by participants | Through study completion, an average of 8 months.
  Measured using a questionnaire
Patients' perception of factors limiting the use of the strategy | Measured at first use of the strategy and at the end of the study follow-up
  Measured using a questionnaire
Healthcare providers' perception of factors limiting the use of the strategy | One and four months after the start of the study
  Measured using a questionnaire
Workload for strategy administrators | Through study completion, an average of 8 months.
  Total time taken by strategy administrators to set up the strategy, explain its functioning to participants and clean it.
Strategy administrators ability to use the strategy | Through study completion, an average of 8 months.
  Measured using a questionnaire
Patients' satisfaction regarding the use of the strategy | Measured at first use of the strategy and at the end of the study follow-up
  Measured using a questionnaire
Healthcare providers' satisfaction regarding the strategy | One and four months after the start of the study
  Measured using a questionnaire
Prevalence of adverse events related to the use of the strategy | Through study completion, an average of 8 months.
  Percentage of times when use of the strategy is stopped early due to adverse events occurring during its use.
Type of adverse events related to the use of the strategy | Through study completion, an average of 8 months.
  Measured using the Simulator Sickness Questionnaire
Severity of adverse events related to the use of the strategy | Through study completion, an average of 8 months.
  Measured using the Simulator Sickness Questionnaire

OTHER OUTCOMES:
Acceptance rate to fill in questionnaires measuring clinical outcomes | Through study completion, an average of 8 months.
  Questionnaires measuring clinical outcomes will include the EORTC Quality of Life Group Core Questionnaire (EORTC QLQ-C30), the State Anxiety Inventory (short form), a visual analogue scale to measure pain, and the Simulator Sickness Questionnaire.
Time taken to fill in questionnaires measuring clinical outcomes | Through study completion, an average of 8 months.
  Questionnaires measuring clinical outcomes will include the EORTC Quality of Life Group Core Questionnaire (EORTC QLQ-C30), the State Anxiety Inventory (short form), a visual analogue scale to measure pain, and the Simulator Sickness Questionnaire.
Completeness of questionnaires measuring clinical outcomes | Through study completion, an average of 8 months.
  Questionnaires measuring clinical outcomes will include the EORTC Quality of Life Group Core Questionnaire (EORTC QLQ-C30), the State Anxiety Inventory (short form), a visual analogue scale to measure pain, and the Simulator Sickness Questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Pauline Boucheron, MD, Principal Investigator — International Agency for Research on Cancer
Locations (1):
- Centre Léon Bérard, Lyon, France

IPD SHARING:
Plan to Share IPD: No